CLINICAL TRIAL: NCT00149643
Title: Fluoxetine for Major Depressive Disorder/Cannabis Disorder in Young People
Brief Title: Effectiveness of Fluoxetine in Young People for the Treatment of Major Depression and Marijuana Dependence
Acronym: CADY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jack Cornelius, Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-19142-1; R01DA019142 (NIH); DPMC
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Depressive Disorder, Major; Cannabis Abuse
Keywords: Cannabis; MDD
MeSH Terms: conditions — Depressive Disorder, Major; Marijuana Abuse | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoxetine (Active Comparator): Gelatin capsules Fluoxetine 10 mg, 1 capsule every a.m. Medication will be increased by one capsule, to a daily dose of fluoxetine 20 mg, 2 capsules barring side effects.
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): Gelatin capsules Placebo capsules, identical to Fluoxetine capsules, 1 capsule every a.m. Medication will be increased by one capsule, to a daily dose of placebo, 2 capsules barring side effects.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fluoxetine — Gelatin capsules Fluoxetine 10 mg, 1 capsule every a.m. Medication will be increased by one capsule, to a daily dose of fluoxetine 20 mg, 2 capsules barring side effects.
  Other Names: Prozac
  Arms: Fluoxetine
Other: Placebo — Gelatin capsules Placebo capsules, identical to Fluoxetine capsules, 1 capsule every a.m. Medication will be increased by one capsule, to a daily dose of placebo, 2 capsules barring side effects.
  Arms: Placebo

SUMMARY:
Adolescents who are diagnosed with major depressive disorder are often also diagnosed with marijuana dependence. Fluoxetine is an antidepressant medication currently used to treat young people who are diagnosed with major depressive disorder. The purpose of this study is to determine the effectiveness of fluoxetine in treating adolescents and young adults diagnosed with both major depressive disorder and marijuana dependence.

DETAILED DESCRIPTION:
Marijuana dependence is the most common illicit substance use disorder in the United States. Its prevalence is highest among adolescents and young adults. Major depressive disorder is one of the most common conditions seen in marijuana dependent individuals. Fluoxetine is an antidepressant medication for treatment of major depression among adolescents and children. The purpose of this study is to determine the effectiveness of fluoxetine in treating adolescents and young people dually diagnosed with major depressive disorder and marijuana dependence.

Participants in this 12-week trial will be randomly assigned to receive either fluoxetine or placebo. Participants will initially be randomly assigned to receive either 10 mg of fluoxetine or placebo. Medication will be given in the morning. If no side effects are observed over the first two weeks of the study, medication will be increased to a daily dose of 20 mg of fluoxetine or placebo. If, at Week 4, a participant continues to demonstrate significant depressive symptoms, medication will be increased to 30 mg daily. All participants will also receive Treatment as Usual (TAU) during the acute phase of the trial, which will consist of motivation enhancement therapy (MET) and Cognitive Behavioral Therapy (CBT). Outcome measures will be obtained at screening, baseline, and weekly intervals for the first four weeks of the treatment phase; they will then be obtained biweekly for the final 8 weeks of the treatment phase. Blood will be drawn at baseline and at Weeks 4, 8, and 12 to assess the level of three liver enzymes (Gamma-glutamyl Transferase (gGTP), Aspartate aminotransferase (SGOT), and Alanine aminotransferase (SGPT)). This will provide a biochemical monitoring of drinking behavior and medication compliance. The 12-week acute phase study will be supplemented by a 9-month naturalistic follow-up phase, during which care will be transferred from the study provider to the community provider. The study will end with a 1-year follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of current marijuana abuse or dependence, confirmed by SCID-SUD
* DSM-IV diagnosis of current major depressive disorder, confirmed by the K-SADS
* Marijuana use of at least two days within the week prior to enrollment
* Demonstrated adequate levels of depressive symptoms within the week prior to enrollment

Exclusion Criteria:

* DSM-IV diagnosis of bipolar disorder, schizoaffective disorder, or schizophrenia
* Hypo or hyperthyroidism
* Significant cardiac, neurological, or kidney impairment
* Liver disease (SGOT, SGPT, or gamma-GTP greater than 3 times the normal level)
* Use of antipsychotic or antidepressant medication in the month prior to enrollment
* DSM-IV dependence on any substance except marijuana or nicotine; alcohol dependence, or history of drug use
* History of significant medication side effects from any SSRI antidepressant
* Pregnant
* Unable to use adequate contraceptive methods for the duration of the study
* Inability to read or understand English

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2004-09; Primary Completion 2009-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack R Cornelius, Principal Investigator — University of Pittsburgh at Pittsburgh
Locations (1):
- Department of Psychiatry, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Cornelius JR, Bukstein OG, Douaihy AB, Clark DB, Chung TA, Daley DC, Wood DS, Brown SJ. Double-blind fluoxetine trial in comorbid MDD-CUD youth and young adults. Drug Alcohol Depend. 2010 Nov 1;112(1-2):39-45. doi: 10.1016/j.drugalcdep.2010.05.010. Epub 2010 Jun 23. PMID 20576364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the Western Psychiatric Institute and Clinic (WPIC) of the University of Pittsburgh Medical Center (UPMC). Subjects were recruited for participation in the treatment study through referrals from any of the WPIC treatment programs and by responding to newspaper, radio, and bus advertisements.
Groups:
- Fluoxetine: Gelatin capsules Fluoxetine 10mg, 1 capsule every a.m. Medication will be increased by one capsule, to a daily dose of fluoxetine 20mg, 2 capsules barring side effects.
- Placebo: Gelatin capsules Placebo capsules,identical to Fluoxetine capsules, 1 capsule every a.m. Medication will be increased by one capsule, to a daily dose of placebo, 2 capsules barring side effects.
Period: Overall Study
Arm/Group | Fluoxetine | Placebo
Started | 34 | 36
Completed | 0 | 0
Not Completed | 34 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoxetine | Placebo | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 32 | 34 | 66
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 21.1 (2.4) | 21.1 (2.4) | 21.1 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 20 | 24 | 44
Region of Enrollment [Number; unit: participants]
  United States | 34 | 36 | 70

OUTCOME MEASURES:

1. Primary Outcome: Days Per Week of Cannabis Use.
Description: The number days out of the last seven days that cannabis was used.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: Days of cannabis use per week
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 34 | 36
Days of cannabis use per week | 3.88 (2.6) | 3.1 (2.27)
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Groups' categorical baseline measures were compared by chi-square analysis, corrected for continuity. Statistical analyses were completed on an intent to-treat study group basis. Outcome measures for depression and for cannabis use and alcohol use across treatment groups were compared by repeated measures analysis of variance. The last observation carried forward (LOCF)method was used for handling missing data in the data analyses; Test type: Superiority or Other; p < 0.05, ANOVA

2. Primary Outcome: Depression Symptoms at Week 12
Description: Average of Beck Depression Inventory (BDI) Scores measured at Weeks 1-4, 6, 8, 10 and 12. The BDI is a subject reported measure that has a minimim score of 0 and a maximum score of 63. A better outcome would consist of values near the minimum end of the scale (0) and a worse outcome would consist of values near the maximum end of the scare (63). Each DSM-IV criteron asses a different depressive symptom.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: BDI Total
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 34 | 36
BDI Total | 7.79 (8.29) | 7.31 (7.98)

3. Secondary Outcome: Number of Cannabis Use Disorder Criterion Met at a Particular Time Point.
Description: Criterion used in this study was the number of DSM-IV cannabis use disorder symptoms (criteria) that were met.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: Number of DSM-IV criterion
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 34 | 36
Number of DSM-IV criterion | 0.59 (0.79) | 0.47 (0.65)

ADVERSE EVENTS:
Time Frame: Adverse events were tracked during the 12-week acute treatment phase.
Arm/Group | Fluoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 0/34 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No